CLINICAL TRIAL: NCT05435014
Title: Phase I/II Randomized, Double-Blind, First-in-Human Study of T-ACE Oil by Trans-Catheter Arterial Embolization or ChemoEmbolization (TAE/TACE) in Patients With Hepatocellular Carcinoma
Brief Title: T-ACE Oil by TAE/TACE in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: T-ACE Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TACE-OHEP-001
Record Dates: First submitted 2021-11-16; First posted 2022-06-28 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ethiodized Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- T-ACE Oil (Experimental): TAE/TACE treatment was performed with T-ACE Oil.
  Interventions: Drug: T-ACE Oil
- Lipiodol (Active Comparator): TAE/TACE treatment was performed with Lipiodol.
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Drug: T-ACE Oil — TAE/TACE treatment was performed with T-ACE Oil. The volume of T-ACE Oil injected would be 1-1.5 mL/cm based on the diameter (cm) of the treated tumor. The maximum dose is 0.25 mL/kg/day but not over 15 mL for each treatment.
  Arms: T-ACE Oil
Drug: Lipiodol — TAE/TACE treatment was performed with Lipiodol. The volume of Lipiodol injected would be 1-1.5 mL/cm based on the diameter (cm) of the treated tumor. The maximum dose is 0.25 mL/kg/day but not over 15 mL for each treatment.
  Arms: Lipiodol

SUMMARY:
The phase I/II, double-blind, randomized study will investigate the efficacy and safety of TACE/TAE treatment with T-ACE Oil in patients with unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Subjects with HCC that meet all eligibility criteria will be admitted to hospital, and TAE or TACE treatment are performed during the hospitalization period; after embolization, subjects are observed in the ward for 1 to 7 days, and evaluated by physician before being discharged. Subjects will be followed up for 7 weeks after treatment for safety and efficacy evaluation.

Phase I part:

12 evaluable subjects will be enrolled sequentially in Phase I part. The first 3 subjects will receive TAE treatment (whether or not they are contraindicated to Doxorubicin) and the following 3 subjects (4th to 6th subjects) will receive TACE treatment. The remaining subjects may receive TAE or TACE treatment. Subjects will be enrolled sequentially in Phase I. For the first six subjects in Phase I, after the subject completes TAE or TACE treatment and is followed for 2 weeks, safety and tolerability data during this period will be reviewed by the safety review committee (SRC); only approved by the SRC, the next subject may start the TAE or TACE treatment. For the 7th to 12th subjects in Phase I, after the subject completes TAE or TACE treatment and is followed until discharge from hospitalization, safety and tolerability data during this period will be reviewed by the safety review committee (SRC); only approved by the SRC, the next subject may start the TAE or TACE treatment. After data for all 12 evaluable subjects are reviewed by SRC and approval is given by the SRC, the study may proceed to Phase II part.

Phase II part:

70 evaluable subjects will be randomized in a 1:1 ratio to receive TAE/TACE treatment by T-ACE Oil or Lipiodol for safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of over 20 years (or according to local legal definition of majority).
2. Patients diagnosed of HCC (Meet at least ONE of the following criteria):

   A. Diagnosed via tumor biopsy by pathologists and confirmed by on-service physician.

   B. High risk patients (viral hepatitis B or C or cirrhotic) with typical liver cancer image appeared on MRI or CT scan.
3. In very early stage to intermediate stage by BCLC staging (2018 AASLD), HCC tumor numbers ≦ 10, HCC tumor size ≦ 15 centimeters (determined by CT, MRI or ultrasound), with liver function at Child-Pugh score[1] ≦ 8.
4. Disease can be treated by trans-arterial chemoembolization, and can be evaluated by Magnetic resonance imaging (MRI), or computed tomography (CT).
5. Patients who only require a single TAE/TACE treatment to treat all HCC tumors at once.
6. Target HCC tumors should have at least 1 tumor that is larger than 1 cm in diameter (determined by CT, MRI or ultrasound) and non-treated before.
7. May have received local therapy such as TAE, TACE, radiofrequency ablation (RFA) or surgery and remain eligible for study provided the prior therapy was within the following timeframes and the subject has fully recovered from prior therapy:

   A. TAE/TACE: more than 8 weeks since completion of prior therapy B. RFA: After PI confirm subject is fully recovered from prior therapy based on screening visit physical examination and liver function laboratory tests results.

   C. Surgery: After PI confirm subject is fully recovered from prior therapy based on screening visit physical examination and liver function laboratory tests results.
8. Patients able to understand, willing to accept and cooperate with all clinical trial practices.
9. Willing to sign a written informed consent form.

Exclusion Criteria:

1. Major branch of portal vein has been invaded by HCC, extrahepatic metastasis or other malignant tumors (current active malignancy or active malignancy within the past 5 years).
2. Eligible for curative surgery or transplant as judged by PI.
3. Evidences of decompensation (Meet at least ONE of the following criteria):

   * Total Bilirubin > 2 mg/dL
   * INR > 1.7
   * Child-Pugh score > 8
   * refractory ascites
   * active bleeding
   * hepatic encephalopathy
   * severe infection
4. Any of the following findings (but not limit to):

   * Heart failure (NYHA Class III or IV), COPD (Stage III or IV).
   * A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Fridericia's QT correction formula.
   * A history of risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or use of concomitant medications that prolong the QT/QTc interval (e.g., class Ia, Ic or III antiarrhythmic drugs, tricyclic antidepressants or phenothiazines)
   * Bronchial asthma that may increase the risk associated with study participation, or may interfere with compliance of the protocol as judged by the PI.
   * Renal dysfunction (eGFR < 50 ml/min/1.73m2 and/or creatinine > 1.5x ULN), or patients is planned to accept any renal replacement therapy during treatment visits.
   * Diagnosed with hyperthyroidism or receiving treatment for hyperthyroidism. Has unstable thyroid function as judged by the PI (e.g. TSH > 5.0 mIU/L).
   * Traumatic injuries, clinically significant hemorrhage/bleeding, or clinically significant gastrointestinal bleeding within 8 weeks.
   * Major cardiovascular disease, including stroke and transient ischemic attack (TIA).
   * Known homocystinuria.
5. Any of the following laboratory findings:

   * Absolute Neutrophil Count < 1000/μL
   * Platelets < 50,000/μL
   * Hgb < 8.5 g/dL
   * AST > 5x ULN
   * ALT > 5x ULN
6. Performance status Eastern Cooperative Oncology Group (ECOG) of 2 or more.
7. Patients whose blood vessel are too difficult to perform TACE procedure as judged by PI.
8. TACE procedure would be performed in areas of the liver where bile ducts are dilated as judged by PI.
9. Prominent Hepatic arteriovenous (AV) shunt, as judged by PI.
10. Non-targeted area may be endangered during TACE procedure, as judged by PI.
11. Patients, who have ever accepted TACE therapy, and cannot gain extra benefits from further embolization treatment.
12. Number of HCC tumors more than 10.
13. Allergy or contraindication to iodine, Lipiodol, allowed contrast agents, allowed Gelfoam suppositories or allowed artery hemostats.
14. Pregnant females or lactating females.
15. Male or female subjects with fertility who are unwilling to perform highly effective contraception method.
16. Subjects who, in the opinion of the investigator, are not suitable to participate in the trial for whatever reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase I part: Incidence of all adverse events (AEs) after TAE/TACE treatment with T-ACE Oil | 7 weeks after treatment
Phase I part: Incidence of adverse events of special interest (AESIs) after TAE/TACE treatment with T-ACE Oil | 7 weeks after treatment
Phase I part: Incidence of all serious adverse events (SAEs) after TAE/TACE treatment with T-ACE Oil | 7 weeks after treatment
Phase I part: Safety variables evaluation - Blood pressures | Pre-intervention (V1)(-28 to -1 days)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - Blood pressures | immediately after the intervention (V2)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - Blood pressures | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - Blood pressures | 2 weeks after treatment (V3)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - Blood pressures | 6 weeks after treatment (V4)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - Blood pressures | 7 weeks after treatment (V5)
  Blood pressures (including SBP and DBP, unit: mmHg)of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | Pre-intervention (V1)(-28 to -1 days)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | immediately after the intervention (V2)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | 2 weeks after treatment (V3)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | 6 weeks after treatment (V4)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - pulse rate | 7 weeks after treatment (V5)
  Pulse rate (beats/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | Pre-intervention (V1)(-28 to -1 days)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | immediately after the intervention (V2)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | 2 weeks after treatment (V3)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | 6 weeks after treatment (V4)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Body weight. | 7 weeks after treatment (V5)
  Body weight (kilograms) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | Pre-intervention (V1)(-28 to -1 days)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | immediately after the intervention (V2)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | 2 weeks after treatment (V3)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | 6 weeks after treatment (V4)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Respiratory rate | 7 weeks after treatment (V5)
  Respiratory rate (times/min) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | Pre-intervention (V1)(-28 to -1 days)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | immediately after the intervention (V2)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | 2 weeks after treatment (V3)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | 6 weeks after treatment (V4)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - Body temperature. | 7 weeks after treatment (V5)
  Body temperature (oC) of subjects will be measured.
Phase I part: Safety variables evaluation - WBC | Pre-intervention (V1)(-28 to -1 days)
  WBC (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - WBC | immediately after the intervention (V2)
  WBC (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - WBC | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  WBC (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - WBC | 2 weeks after treatment (V3)
  WBC (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - WBC | 6 weeks after treatment (V4)
  WBC (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Platelet count | Pre-intervention (V1)(-28 to -1 days)
  Platelet count (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Platelet count | immediately after the intervention (V2)
  Platelet count (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Platelet count | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Platelet count (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Platelet count | 2 weeks after treatment (V3)
  Platelet count (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Platelet count | 6 weeks after treatment (V4)
  Platelet count (1000/uL) of subjects will be measured.
Phase I part: Safety variables evaluation - Hb | Pre-intervention (V1)(-28 to -1 days)
  Hb (g/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Hb | immediately after the intervention (V2)
  Hb (g/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Hb | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Hb (g/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Hb | 2 weeks after treatment (V3)
  Hb (g/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Hb | 6 weeks after treatment (V4)
  Hb (g/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - blood urea nitrogen test | Pre-intervention (V1)(-28 to -1 days)
  BUN (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - blood urea nitrogen test | immediately after the intervention (V2)
  BUN (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - blood urea nitrogen test | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  BUN (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - blood urea nitrogen test | 2 weeks after treatment (V3)
  BUN (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - blood urea nitrogen test | 6 weeks after treatment (V4)
  BUN (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Bilirubin | Pre-intervention (V1)(-28 to -1 days)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Bilirubin | immediately after the intervention (V2)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Bilirubin | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Bilirubin | 2 weeks after treatment (V3)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Bilirubin | 6 weeks after treatment (V4)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Renal function | Pre-intervention (V1)(-28 to -1 days)
  Creatinine (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Renal function | immediately after the intervention (V2)
  Creatinine (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Renal function | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Creatinine (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Renal function | 2 weeks after treatment (V3)
  Creatinine (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Renal function | 6 weeks after treatment (V4)
  Creatinine (mg/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Liver function | Pre-intervention (V1)(-28 to -1 days)
  AST and ALT (U/L) of subjects will be measured.
Phase I part: Safety variables evaluation - Liver function | immediately after the intervention (V2)
  AST and ALT (U/L) of subjects will be measured.
Phase I part: Safety variables evaluation - Liver function | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  AST and ALT (U/L) of subjects will be measured.
Phase I part: Safety variables evaluation - Liver function | 2 weeks after treatment (V3)
  AST and ALT (U/L) of subjects will be measured.
Phase I part: Safety variables evaluation - Liver function | 6 weeks after treatment (V4)
  AST and ALT (U/L) of subjects will be measured.
Phase I part: Safety variables evaluation - Coagulation function | Pre-intervention (V1)(-28 to -1 days)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase I part: Safety variables evaluation - Coagulation function | immediately after the intervention (V2)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase I part: Safety variables evaluation - Coagulation function | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase I part: Safety variables evaluation - Coagulation function | 2 weeks after treatment (V3)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase I part: Safety variables evaluation - Coagulation function | 6 weeks after treatment (V4)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (T3) | Pre-intervention (V1)(-28 to -1 days)
  T3 (ng/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (T3) | 6 weeks after treatment (V4).
  T3 (ng/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (Free T4) | Pre-intervention (V1)(-28 to -1 days)
  T4 (ng/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (Free T4) | 6 weeks after treatment (V4).
  T4 (ng/dL) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (TSH) | Pre-intervention (V1)(-28 to -1 days)
  TSH (uIU/ml) of subjects will be measured.
Phase I part: Safety variables evaluation - Thyroid function (TSH) | 6 weeks after treatment (V4).
  TSH (uIU/ml) of subjects will be measured.
Phase I part: Safety variables evaluation - ECG test | Pre-intervention (V1)(-28 to -1 days)
  Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0
Phase I part: Safety variables evaluation - ECG test | immediately after the intervention (V2)
  Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0
Phase I part: Safety variables evaluation - ECG test | 6 weeks after treatment (V4)
  Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0
Phase II part: T-ACE Oil or Lipiodol deposition type on CT scan after TAE/TACE treatment. | 72 hours after treatment
  CT or MRI image should be taken at the screening visit, after the TAE or TACE procedure and visit 4 (6 weeks after TAE or TACE procedure). No additional contrast will be administered for the CT after TAE or TACE procedure. V1 and V4 image evaluation will be performed by MRI. V2 image evaluation method will be performed by CT scan. If the subject has had an MRI examination within 28 days before TAE/TACE treatment, the V1 MRI can be skipped.
Phase II part: mRECIST overall response at 6 weeks after TAE/TACE treatment. | 6 weeks after treatment.
  mRECIST (modified Response Evaluation Criteria in Solid Tumors) overall response and mRECIST target lesion response will be evaluated based on the image taken at the screening visit and at visit 4 (6 weeks after TAE or TACE procedure). mRECIST overall response for each patient will be categorized: Complete response (CR), Partial response (PR), Stable disease (SD), and Progressive disease (PD). mRECIST overall response is based on target lesions and non-target lesions responses and appearance of new lesions and/or extra-hepatic disease.
Phase II part: target lesion response at 6 weeks after TAE/TACE treatment. | 6 weeks after treatment.
  target lesion response will be evaluated based on the image

SECONDARY OUTCOMES:
Phase I part: T-ACE Oil deposition type on CT scan after TAE/TACE treatment with T-ACE Oil. | 72 hours after treatment
  CT or MRI image should be taken at the screening visit, after the TAE or TACE procedure and visit 4 (6 weeks after TAE or TACE procedure). No additional contrast will be administered for the CT after TAE or TACE procedure. V1 and V4 image evaluation will be performed by MRI. V2 image evaluation method will be performed by CT scan. If the subject has had an MRI examination within 28 days before TAE/TACE treatment, the V1 MRI can be skipped.
Phase I part: mRECIST overall response at 6 weeks after TAE/TACE treatment with T-ACE Oil. | 6 weeks after treatment.
  mRECIST (modified Response Evaluation Criteria in Solid Tumors) overall response and mRECIST target lesion response will be evaluated based on the image taken at the screening visit and at visit 4 (6 weeks after TAE or TACE procedure). mRECIST overall response for each patient will be categorized: Complete response (CR), Partial response (PR), Stable disease (SD), and Progressive disease (PD). mRECIST overall response is based on target lesions and non-target lesions responses and appearance of new lesions and/or extra-hepatic disease.
Phase I part: target lesion response at 6 weeks after TAE/TACE treatment with T-ACE Oil. | 6 weeks after treatment.
  target lesion response will be evaluated based on the image
Phase II part: Incidence of all adverse events (AEs) after TAE/TACE treatment with T-ACE Oil or Lipiodol. | 7 weeks after treatment
Phase II part: Incidence of adverse events of special interest (AESIs) after TAE/TACE treatment with T-ACE Oil or Lipiodol. | 7 weeks after treatment
Phase II part: Incidence of all serious adverse events (SAEs) after TAE/TACE treatment with T-ACE Oil or Lipiodol. | 7 weeks after treatment
Phase II part: Safety variables evaluation - Blood pressures | Pre-intervention (V1)(-28 to -1 days)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Blood pressures | immediately after the intervention (V2)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Blood pressures | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Blood pressures | 2 weeks after treatment (V3)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Blood pressures | 6 weeks after treatment (V4)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Blood pressures | 7 weeks after treatment (V5)
  Blood pressures (including SBP and DBP, unit: mmHg) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | Pre-intervention (V1)(-28 to -1 days)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | immediately after the intervention (V2)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | 2 weeks after treatment (V3)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | 6 weeks after treatment (V4)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Pulse rate | 7 weeks after treatment (V5)
  Pulse rate (beats/min) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | Pre-intervention (V1)(-28 to -1 days)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | immediately after the intervention (V2)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | 2 weeks after treatment (V3)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | 6 weeks after treatment (V4)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body weight. | 7 weeks after treatment (V5)
  Body weight (kilograms) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | Pre-intervention (V1)(-28 to -1 days)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | immediately after the intervention (V2)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | 2 weeks after treatment (V3)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | 6 weeks after treatment (V4)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - Body temperature. | 7 weeks after treatment (V5)
  Body temperature (oC) of subjects will be measured.
Phase II part: Safety variables evaluation - WBC | Pre-intervention (V1)(-28 to -1 days)
  WBC (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - WBC | immediately after the intervention (V2)
  WBC (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - WBC | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  WBC (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - WBC | 2 weeks after treatment (V3)
  WBC (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - WBC | 6 weeks after treatment (V4)
  WBC (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Platelet count | Pre-intervention (V1)(-28 to -1 days)
  Platelet count (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Platelet count | immediately after the intervention (V2)
  Platelet count (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Platelet count | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Platelet count (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Platelet count | 2 weeks after treatment (V3)
  Platelet count (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Platelet count | 6 weeks after treatment (V4)
  Platelet count (1000/uL) of subjects will be measured.
Phase II part: Safety variables evaluation - Hb | Pre-intervention (V1)(-28 to -1 days)
  Hb (g/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Hb | immediately after the intervention (V2)
  Hb (g/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Hb | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Hb (g/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Hb | 2 weeks after treatment (V3)
  Hb (g/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Hb | 6 weeks after treatment (V4)
  Hb (g/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - blood urea nitrogen test | Pre-intervention (V1)(-28 to -1 days)
  BUN (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - blood urea nitrogen test | immediately after the intervention (V2)
  BUN (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - blood urea nitrogen test | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  BUN (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - blood urea nitrogen test | 2 weeks after treatment (V3)
  BUN (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - blood urea nitrogen test | 6 weeks after treatment (V4)
  BUN (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Bilirubin | Pre-intervention (V1)(-28 to -1 days)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Bilirubin | immediately after the intervention (V2)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Bilirubin | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Bilirubin | 2 weeks after treatment (V3)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Bilirubin | 6 weeks after treatment (V4)
  Bilirubin-T and Bilirubin-D (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Renal function | Pre-intervention (V1)(-28 to -1 days)
  Creatinine (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Renal function | immediately after the intervention (V2)
  Creatinine (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Renal function | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Creatinine (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Renal function | 2 weeks after treatment (V3)
  Creatinine (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Renal function | 6 weeks after treatment (V4)
  Creatinine (mg/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Liver function | Pre-intervention (V1)(-28 to -1 days)
  AST and ALT (U/L) of subjects will be measured.
Phase II part: Safety variables evaluation - Liver function | 6 weeks after treatment (V4)
  AST and ALT (U/L) of subjects will be measured.
Phase II part: Safety variables evaluation - Coagulation function | Pre-intervention (V1)(-28 to -1 days)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase II part: Safety variables evaluation - Coagulation function | immediately after the intervention (V2)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase II part: Safety variables evaluation - Coagulation function | discharge of hospitalization (V2A)(1 to 7 days of discharge of hospitalization)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase II part: Safety variables evaluation - Coagulation function | 2 weeks after treatment (V3)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase II part: Safety variables evaluation - Coagulation function | 6 weeks after treatment (V4)
  Prothrombin time and APTT (seconds) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (T3) | Pre-intervention (V1)(-28 to -1 days)
  T3 (ng/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (T3) | 6 weeks after treatment (V4)
  T3 (ng/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (Free T4) | Pre-intervention (V1)(-28 to -1 days)
  T4 (ng/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (Free T4) | 6 weeks after treatment (V4)
  T4 (ng/dL) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (TSH) | Pre-intervention (V1)(-28 to -1 days)
  TSH (uIU/ml) of subjects will be measured.
Phase II part: Safety variables evaluation - Thyroid function (TSH) | 6 weeks after treatment (V4)
  TSH (uIU/ml) of subjects will be measured.
Phase II part: Safety variables evaluation - ECG test | Pre-intervention (V1)(-28 to -1 days)
  each component of Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0
Phase II part: Safety variables evaluation - ECG test | immediately after the intervention (V2)
  each component of Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0
Phase II part: Safety variables evaluation - ECG test | 6 weeks after treatment (V4)
  each component of Electrocardiogram (ECG) of subjects will be measured. The participants with treatment-related adverse events will be assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chin Liang, PhD, MD, Principal Investigator — National Taiwan University Hospital; Xi-Zhang Lin, MD, Study Chair — T-ACE Medical Co., Ltd
Locations (4):
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Tungs' Taichung Metroharbor Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Background] Miyayama S, Yamashiro M, Okuda M, Yoshie Y, Sugimori N, Igarashi S, Nakashima Y, Notsumata K, Toya D, Tanaka N, Mitsui T, Matsui O. Chemoembolization for the treatment of large hepatocellular carcinoma. J Vasc Interv Radiol. 2010 Aug;21(8):1226-34. doi: 10.1016/j.jvir.2010.04.015. Epub 2010 Jul 3. PMID 20598571
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] Lencioni R, de Baere T, Soulen MC, Rilling WS, Geschwind JF. Lipiodol transarterial chemoembolization for hepatocellular carcinoma: A systematic review of efficacy and safety data. Hepatology. 2016 Jul;64(1):106-16. doi: 10.1002/hep.28453. Epub 2016 Mar 7. PMID 26765068
- [Background] Wang Z, Lin M, Lesage D, Chen R, Chapiro J, Gu T, Tacher V, Duran R, Geschwind JF. Three-dimensional evaluation of lipiodol retention in HCC after chemoembolization: a quantitative comparison between CBCT and MDCT. Acad Radiol. 2014 Mar;21(3):393-9. doi: 10.1016/j.acra.2013.11.006. PMID 24507426